CLINICAL TRIAL: NCT00730405
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-ranging Study to Investigate the Efficacy and Safety of 4 Dose Regimens of Oral Albaconazole in Subjects With Distal Subungual Onychomycosis
Brief Title: Efficacy and Safety Study of 4 Dose Regimens of Oral Albaconazole in Subjects With Distal Subungual Onychomycosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114554
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-01

CONDITIONS: Onychomycosis
Keywords: Distal, Subungual onychomycosis; onychomycosis; nail fungus; Toenail fungus
MeSH Terms: conditions — Onychomycosis | interventions — albaconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Albaconazole 100mg (Active Comparator): Albaconazole for 36 weeks
  Interventions: Drug: Albaconazole 100mg
- Albaconazole 200mg (Active Comparator): Albaconazole for 36 weeks
  Interventions: Drug: Albaconazole 200mg
- Albaconazole 400mg (Active Comparator): Albaconazole for 36 weeks
  Interventions: Drug: Albaconazole 400mg
- Albaconazole 400mg 24 weeks, Placebo 12 weeks (Active Comparator): Albaconazole for 24 weeks, Placebo for 12 weeks
  Interventions: Drug: Albaconazole 400mg; Drug: Placebo 400 mg
- Placebo 400 mg (Placebo Comparator): Placebo for 36 weeks
  Interventions: Drug: Placebo 400 mg

INTERVENTIONS:
Drug: Albaconazole 100mg — Albaconazole for 36 weeks
  Arms: Albaconazole 100mg
Drug: Albaconazole 200mg — Albaconazole for 36 weeks
  Arms: Albaconazole 200mg
Drug: Albaconazole 400mg — Albaconazole for 36 weeks
  Arms: Albaconazole 400mg
Drug: Albaconazole 400mg — Albaconazole for 24 weeks, Placebo for 12 weeks
  Arms: Albaconazole 400mg 24 weeks, Placebo 12 weeks
Drug: Placebo 400 mg — Placebo for 36 weeks
  Arms: Albaconazole 400mg 24 weeks, Placebo 12 weeks; Placebo 400 mg

SUMMARY:
Phase 2 study to examine how the study drug works and its side effects in subjects with toenail fungus.

DETAILED DESCRIPTION:
A phase 2, randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study to investigate the efficacy and safety of 4 dose regimens of ORAL albaconazole in subjects with distal subungual onychomycosis. Subjects will take oral study drug for up to 36 weeks and then will be followed for an additional 16 weeks to determine if the study drug was efficacious. Subjects will have routine blood draws and other safety assessments during the study, as well as regular assessments of their toenail fungus

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 to 75 years.
* Diagnosis with distal subungual onychomycosis of the toenails that affects at least one great toe (target toenail).
* Subject is willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol-specific procedures are performed.
* Subject is able to complete the study, comply with study instructions, and take study product orally.
* Sexually active non-lactating females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception while receiving protocol-assigned product and up to the first menses 60 days following the last dose of study product.
* Women of childbearing potential must have a negative pregnancy test at enrollment.
* Subject has screening laboratory parameters and ECG within the normal ranges unless considered to be not clinically relevant by the principal investigator.

Exclusion Criteria:

Subjects with any of the following conditions or characteristics will be excluded from study enrollment (ie, will not receive study product):

* Subject has received an investigational drug within 4 weeks of the first dose of study product, or who are scheduled to receive an investigational drug other than the study product during the study.
* Subject has participated in a clinical trial for the systemic treatment of onychomycosis of the toenails within 6 months prior to the first dose of study product.
* Subject is receiving any drugs that are known substrates of the 3A4 isozyme of cytochrome P450 (CYP3A4) with QT prolongation potential or any of the concomitant medications listed under prohibited medication section.
* Subject has a history of known or suspected intolerance to albaconazole or the formulation excipients, or to azole antifungal drugs in general.
* Subject has previously participated in a clinical study with albaconazole.
* Subject is not prepared to give up use of any nail cosmetic products for the duration of the study.
* Subject has any known immunodeficiency or history of malignancy in the last 4 years, excluding nonmelanoma skin cancer.
* Subject has any known liver disease or a history of liver toxicity with other drugs.
* Subject is currently suffering from any disease or condition, that could include abnormal laboratory tests, and/or who are currently using medication which in the opinion of the investigator may affect the evaluation of the study product or place the subject at undue risk.
* Subject has psoriasis, lichen planus, or other abnormalities that could result in a clinically abnormal toenail.
* Subject has a history of any condition that could possibly affect absorption of drug (eg, gastrectomy), uncontrolled diabetes, clinically significant peripheral vascular disease or peripheral circulatory impairment, or has had any major illness within 30 days prior to the screening examination.
* Subject has a history of drug, prescription medicine, or alcohol abuse within the past 2 years.
* Female subjects who are pregnant, trying to become pregnant, or lactating.
* Employees of Investigator/clinical research organization (CRO) or Stiefel Laboratories, Inc., or an immediate family member (partner, offspring, parents, siblings or sibling's offspring) of an employee.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2008-07-16 (Actual); Primary Completion 2010-02-19 (Actual); Study Completion 2010-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (33):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Genova Clinical Research, Tucson, Arizona
  - Impact Clinical Trials, Beverly Hills, California
  - Northern California Research, Carmichael, California
  - Center for Dermatology Clinical Research, Fremont, California
  - Therapeutics Clinical Research, San Diego, California
  - UCSF Dermatology Research, San Francisco, California
  - Thomas J. Stephens & Associates, Inc. Colorado Research Center, Colorado Springs, Colorado
  - International Dermatology Research Inc, Miami, Florida
  - Greater Miami Skin & Laser Center, Miami Beach, Florida
  - Miami Dermatology Research Institute LLC, North Miami Beach, Florida
  - MedaPhase, Inc, Newnan, Georgia
  - Gwinnett Clinical Research Center, Inc., Snellville, Georgia
  - Welborn Clinic, Evansville, Indiana
  - Henry Ford Medical Center, Detroit, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Skin Specialists, Inc, Omaha, Nebraska
  - NYU Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oregon Dermatology & Research Centre, Portland, Oregon
  - Oregon Medical, Portland, Oregon
  - The Skin Wellness Center, Knoxville, Tennessee
  - Tennessee Clinical Research, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - J & S Studies, Inc., College Station, Texas
  - Research Across America, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - DermatologyResearch Center, Salt Lake City, Utah
  - Education and Research Foundation, Lynchburg, Virginia
- Canada (3):
  - Ultranova Skincare, Barrie, Ontario
  - North Bay Dermatology Centre Inc., North Bay, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario
- Dermatology Centre, University of Iceland, Hudlaeknaslodin, Kopavogur, Iceland

REFERENCES:
- [Background] Sigurgeirsson B, van Rossem K, Malahias S, Raterink K. A phase II, randomized, double-blind, placebo-controlled, parallel group, dose-ranging study to investigate the efficacy and safety of 4 dose regimens of oral albaconazole in patients with distal subungual onychomycosis. J Am Acad Dermatol. 2013 Sep;69(3):416-25. doi: 10.1016/j.jaad.2013.03.021. Epub 2013 May 22. PMID 23706639
- See also: Results for study 114554 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/114554?search=study&search_terms=114554#rs

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 16 July 2008 to 19 February 2010, total of 582 participants with onychomycosis were randomized in 5 different arms at 26 centres in the United States, 3 centres in the Canada and 1 centre in the Iceland.
Groups:
- Albaconazole 400 mg (36 Weeks) Oral Weekly: Participants received 4 capsules containing 100 milligrams (mg) of albaconazole in combination with amino methacrylate copolymer as film coated microcrystalline cellulose spheres once every week for 36 weeks. Albaconazole film-coated spheres are filled in size 1, off white, hard gelatin capsules. The capsules were swallowed whole with water, not chewed or crushed. Study product was administered every 7 days. Visits were scheduled on dosing days; dosing on visit dates was administered at the site.
- Albaconazole 400 mg (24 Weeks) Oral Weekly: Participants received 4 capsules containing 100 mg of albaconazole in combination with amino methacrylate copolymer as film coated microcrystalline cellulose spheres once every week for 24 weeks followed by 4 placebo capsules every week for 12 weeks. Albaconazole film-coated spheres are filled in size 1, off white, hard gelatin capsules. Placebo capsules with identical ingredients and packaging as albaconazole capsules but without the active ingredient albaconazole. The capsules were swallowed whole with water, not chewed or crushed. Study product was administered every 7 days. Visits were scheduled on dosing days; dosing on visit dates was administered at the site.
- Albaconazole 200 mg (36 Weeks) Oral Weekly: Participants received 4 capsules (2 active + 2 placebo) containing 100 mg of albaconazole in combination with amino methacrylate copolymer as film coated microcrystalline cellulose spheres once every week for 36 weeks. Albaconazole film-coated spheres are filled in size 1, off white, hard gelatin capsules. Placebo capsules with identical ingredients and packaging as albaconazole capsules but without the active ingredient albaconazole. The capsules were swallowed whole with water, not chewed or crushed. Study product was administered every 7 days. Visits were scheduled on dosing days; dosing on visit dates was administered at the site.
- Albaconazole 100 mg (36 Weeks) Oral Weekly: Participants received 4 capsules (1 active + 3 placebo) containing 100 mg of albaconazole in combination with amino methacrylate copolymer as film coated microcrystalline cellulose spheres once every week for 36 weeks. Albaconazole film-coated spheres are filled in size 1, off white, hard gelatin capsules. Placebo capsules with identical ingredients and packaging as albaconazole capsules but without the active ingredient albaconazole. The capsules were swallowed whole with water, not chewed or crushed. Study product was administered every 7 days. Visits were scheduled on dosing days; dosing on visit dates was administered at the site.
- Placebo: Participants received 4 placebo capsules with identical ingredients and packaging as albaconazole capsules but without the active ingredient albaconazole. The capsules were swallowed whole with water, not chewed or crushed. Study product was administered every 7 days. Visits were scheduled on dosing days; dosing on visit dates was administered at the site.
Period: Overall Study-Treatment Phase
Arm/Group | Albaconazole 400 mg (36 Weeks) Oral Weekly | Albaconazole 400 mg (24 Weeks) Oral Weekly | Albaconazole 200 mg (36 Weeks) Oral Weekly | Albaconazole 100 mg (36 Weeks) Oral Weekly | Placebo
Started | 116 | 117 | 117 | 117 | 115
Completed | 97 | 96 | 96 | 98 | 95
Not Completed | 19 | 21 | 21 | 19 | 20
Not completed — Adverse Event | 5 | 10 | 4 | 8 | 4
Not completed — Lost to Follow-up | 4 | 5 | 6 | 4 | 4
Not completed — Non-compliance with Study Treatment | 1 | 0 | 5 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 1 | 2 | 5 | 8
Not completed — Did not met eligibility | 0 | 0 | 1 | 0 | 0
Not completed — Participant meets exclusion | 0 | 0 | 1 | 0 | 0
Not completed — Prohibited concomitant medication | 1 | 0 | 0 | 0 | 0
Not completed — Withdrew from study treatment | 0 | 1 | 0 | 0 | 0
Not completed — Use of prohibited medication | 0 | 1 | 0 | 0 | 2
Not completed — Human immunodeficiency virus positive | 0 | 0 | 1 | 0 | 0
Not completed — Misrandomized | 0 | 1 | 0 | 0 | 0
Not completed — Study drug interrupted | 0 | 1 | 0 | 0 | 0
Not completed — Due to in-vitro fertilization | 0 | 0 | 0 | 1 | 0
Not completed — Protocol violation due to eligibility | 0 | 0 | 1 | 0 | 0
Not completed — Change of location | 0 | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0
Not completed — QTCF: 454 millisecond, withdrew consent | 0 | 0 | 0 | 0 | 1
Not completed — Atrial fibrillation history | 1 | 0 | 0 | 0 | 0
Period: Overall Study-follow-up Phase
Arm/Group | Albaconazole 400 mg (36 Weeks) Oral Weekly | Albaconazole 400 mg (24 Weeks) Oral Weekly | Albaconazole 200 mg (36 Weeks) Oral Weekly | Albaconazole 100 mg (36 Weeks) Oral Weekly | Placebo
Started | 116 | 117 | 117 | 117 | 115
Completed | 95 | 96 | 94 | 100 | 93
Not Completed | 21 | 21 | 23 | 17 | 22
Not completed — Adverse Event | 2 | 6 | 2 | 3 | 4
Not completed — Lost to Follow-up | 7 | 6 | 8 | 4 | 6
Not completed — Withdrawal by Subject | 7 | 3 | 3 | 6 | 10
Not completed — Death | 0 | 1 | 0 | 1 | 0
Not completed — Change of location | 1 | 1 | 0 | 1 | 0
Not completed — Did not met eligibility | 0 | 0 | 1 | 0 | 0
Not completed — Non-compliance with study treatment | 0 | 0 | 1 | 0 | 0
Not completed — Participant meets exclusion criteria | 0 | 0 | 1 | 0 | 0
Not completed — Terminated due to adverse event (AE) | 0 | 0 | 0 | 0 | 1
Not completed — Prohibited concomitant medication | 1 | 0 | 0 | 0 | 0
Not completed — Refused follow-up due to AE | 0 | 0 | 0 | 1 | 0
Not completed — Requested to withdraw from follow-up | 0 | 1 | 1 | 0 | 0
Not completed — Declined to continue with follow-up | 1 | 1 | 0 | 0 | 0
Not completed — Use of restricted medication | 0 | 1 | 0 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 2 | 0 | 0
Not completed — Missing | 0 | 0 | 2 | 0 | 0
Not completed — Use an exclusionary medication | 0 | 0 | 0 | 0 | 1
Not completed — Human immunodeficiency virus positive | 0 | 0 | 1 | 0 | 0
Not completed — Mis-randomized | 0 | 1 | 0 | 0 | 0
Not completed — Other Protocol violation | 0 | 0 | 1 | 0 | 0
Not completed — discontinued AE, investigator discretion | 0 | 0 | 0 | 1 | 0
Not completed — Atrial fibrillation history | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Albaconazole 400 mg (36 Weeks) Oral Weekly: Participants received 4 capsules containing 100 mg of albaconazole in combination with amino methacrylate copolymer as film coated microcrystalline cellulose spheres once every week for 36 weeks. Albaconazole film-coated spheres are filled in size 1, off white, hard gelatin capsules. The capsules were swallowed whole with water, not chewed or crushed. Study product was administered every 7 days. Visits were scheduled on dosing days; dosing on visit dates was administered at the site.
- Total: Total of all reporting groups
Arm/Group | Albaconazole 400 mg (36 Weeks) Oral Weekly | Albaconazole 400 mg (24 Weeks) Oral Weekly | Albaconazole 200 mg (36 Weeks) Oral Weekly | Albaconazole 100 mg (36 Weeks) Oral Weekly | Placebo | Total
Number analyzed (Participants) | 116 | 117 | 117 | 117 | 115 | 582
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (11.4) | 49.2 (12.4) | 49.0 (11.0) | 46.8 (12.3) | 48.5 (12.3) | 48.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 23 | 33 | 32 | 141
  Male | 88 | 92 | 94 | 84 | 83 | 441
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 1 | 0 | 4
  Asian | 3 | 3 | 1 | 2 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1 | 2
  Black or African American | 14 | 16 | 7 | 16 | 13 | 66
  White | 95 | 92 | 105 | 93 | 96 | 481
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 4 | 5 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Who Achieve Effective Treatment at Week 52
Description: At each study visit, the investigator assessed the percentage of affected toenail on the target nail by estimating the percent affected nail in each quadrant, summing the percent affected in each quadrant and dividing the sum by 4. Effective treatment was defined as a mycological cure and clear or almost clear nail (distal subungual hyperkeratosis and/or onycholysis leaving less than 10% of nail plate effected). Comparisons were carried out in a sequential step-down fashion, combined with the Holm procedure at step 2. P-value was based on a sequential step-down combined with the Holm procedure. It was assessed on Week 4, 8, 12, 16, 20, 24, 30, 36, 44 and 52.
Time Frame: Week 52
Population: The intent-to-treat (ITT) analysis set consists of all randomized participants who receive study product. All participants were available at the time of assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Albaconazole 400 mg (36 Weeks) Oral Weekly | Albaconazole 400 mg (24 Weeks) Oral Weekly | Albaconazole 200 mg (36 Weeks) Oral Weekly | Albaconazole 100 mg (36 Weeks) Oral Weekly | Placebo
Number analyzed (Participants) | 116 | 117 | 117 | 117 | 115
Percentage of participants | 54 [45.2 to 63.4] | 38 [28.8 to 46.4] | 29 [20.8 to 37.3] | 21 [13.2 to 27.8] | 1 [0.0 to 2.6]
Statistical Analysis 1: Comparison: Albaconazole 400 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Albaconazole 400 mg (24 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Albaconazole 200 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Albaconazole 100 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: The Percentage of Participants Who Achieve Clinical Cure at Week 52
Description: At each study visit, the investigator assessed the percentage of affected toenail on the target nail by estimating the percent affected nail in each quadrant, summing the percent affected in each quadrant and dividing the sum by 4. Clinical cure was defined as 100% clear nail. It was assessed on Week 4, 8, 12, 16, 20, 24, 30, 36, 44 and 52.
Time Frame: Week 52
Population: ITT analysis set. All participants were available at the time of assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Albaconazole 400 mg (36 Weeks) Oral Weekly; Placebo: Participants received 4 placebo capsules with identical ingredients and packaging as albaconazole capsules but without the active ingredient albaconazole. The capsules were swallowed whole with water, not chewed or crushed. Study product was administered every 7 days. Visits were scheduled on dosing days; dosing on visit dates was administered at the site.
Arm/Group | Albaconazole 400 mg (36 Weeks) Oral Weekly | Albaconazole 400 mg (24 Weeks) Oral Weekly | Albaconazole 200 mg (36 Weeks) Oral Weekly | Albaconazole 100 mg (36 Weeks) Oral Weekly | Placebo
Number analyzed (Participants) | 116 | 117 | 117 | 117 | 115
Percentage of participants | 34 [25.0 to 42.2] | 32 [23.2 to 40.0] | 30 [21.6 to 38.2] | 16 [9.6 to 22.9] | 1 [0.0 to 2.6]
Statistical Analysis 1: Comparison: Albaconazole 400 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Albaconazole 400 mg (24 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Albaconazole 200 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Albaconazole 100 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

3. Secondary Outcome: The Percentage of Participants Who Achieve Mycological Cure at Week 52
Description: At each study visit, the investigator assessed the percentage of affected toenail on the target nail by estimating the percent affected nail in each quadrant, summing the percent affected in each quadrant and dividing the sum by 4. Mycological cure was defined as negative potassium hydroxide (KOH) and negative cultures for dermatophytes. It was assessed on Week 12, 16, 20, 24, 30, 36, 44 and 52.
Time Frame: Week 52
Population: ITT analysis set. All participants were available at the time of assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Albaconazole 400 mg (24 Weeks) Oral Weekly: Participants received 4 capsules containing 100 mg of albaconazole in combination with amino methacrylate copolymer as film coated microcrystalline cellulose spheres once every week for 36 weeks. Albaconazole film-coated spheres are filled in size 1, off white, hard gelatin capsules. The capsules were swallowed whole with water, not chewed or crushed. Study product was administered every 7 days. Visits were scheduled on dosing days; dosing on visit dates was administered at the site.
Arm/Group | Albaconazole 400 mg (36 Weeks) Oral Weekly | Albaconazole 400 mg (24 Weeks) Oral Weekly | Albaconazole 200 mg (36 Weeks) Oral Weekly | Albaconazole 100 mg (36 Weeks) Oral Weekly | Placebo
Number analyzed (Participants) | 116 | 117 | 117 | 117 | 115
Percentage of participants | 71 [62.4 to 79.0] | 54 [44.8 to 62.9] | 43 [33.8 to 51.7] | 34 [25.6 to 42.8] | 6 [1.7 to 10.5]
Statistical Analysis 1: Comparison: Albaconazole 400 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Albaconazole 400 mg (24 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Albaconazole 200 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Albaconazole 100 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

4. Secondary Outcome: The Percentage of Participants Who Achieve Complete Cure at Week 52
Description: At each study visit, the investigator assessed the percentage of affected toenail on the target nail by estimating the percent affected nail in each quadrant, summing the percent affected in each quadrant and dividing the sum by 4. Complete cure was defined as mycological cure plus clinical cure. It was assessed on Week 4, 8, 12, 16, 20, 24, 30, 36, 44 and 52.
Time Frame: Week 52
Population: ITT analysis set. All participants were available at the time of assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Albaconazole 400 mg (36 Weeks) Oral Weekly | Albaconazole 400 mg (24 Weeks) Oral Weekly | Albaconazole 200 mg (36 Weeks) Oral Weekly | Albaconazole 100 mg (36 Weeks) Oral Weekly | Placebo
Number analyzed (Participants) | 116 | 117 | 117 | 117 | 115
Percentage of participants | 33 [24.2 to 41.3] | 26 [17.7 to 33.6] | 21 [13.2 to 27.8] | 12 [6.1 to 17.8] | 0 [NA to NA] — 95% confidence interval not derived, as no participant achieved complete response.
Statistical Analysis 1: Comparison: Albaconazole 400 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Albaconazole 400 mg (24 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Albaconazole 200 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Albaconazole 100 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

5. Secondary Outcome: Absolute Change in Unaffected Part of Target Nail From Baseline to Week 52
Description: Length of the unaffected part of the target nail was measured in millimeters along the midpoint from the nail fold to the proximal border of the affected part (lowest point affected) along the midpoint of the target nail. It was assessed on Week 4, 8, 12, 16, 20, 24, 30, 36, 44 and 52. Baseline values were the observations at Week 0/Day 1 or before. Change from Baseline was a Baseline value subtracted from Week 52 value. P-value was based on analysis of variance (ANOVA) with treatment and pooled center. Statistics is provided for adjusted least square mean.
Time Frame: Baseline (Week 0/Day 1 or before) and up to Week 52
Population: ITT analysis set. All participants were available at the time of assessment.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Albaconazole 400 mg (36 Weeks) Oral Weekly | Albaconazole 400 mg (24 Weeks) Oral Weekly | Albaconazole 200 mg (36 Weeks) Oral Weekly | Albaconazole 100 mg (36 Weeks) Oral Weekly | Placebo
Number analyzed (Participants) | 116 | 117 | 117 | 117 | 115
Millimeters | 6.47 (4.62) | 6.21 (4.51) | 4.75 (4.58) | 3.78 (4.94) | 0.40 (3.14)
Statistical Analysis 1: Comparison: Albaconazole 400 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Net) = -6.10, Standard Error of Mean 0.57
Statistical Analysis 2: Comparison: Albaconazole 400 mg (24 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Net) = -5.71, Standard Error of Mean 0.57
Statistical Analysis 3: Comparison: Albaconazole 200 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Net) = -4.44, Standard Error of Mean 0.57
Statistical Analysis 4: Comparison: Albaconazole 100 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Mean Difference (Net) = -3.22, Standard Error of Mean 0.58

6. Secondary Outcome: The Percentage of Participants With a Global Change Score of Cleared or Much Improved at Week 52
Description: A count of the number of toenails affected, using visual examination, was performed at all study visits (Week 12, 24, 30, 36, 44 and 52). The investigator given a global evaluation of the toenails condition, based on the investigator's assessment of the reduction in extent of nail involvement and improvement in clinical signs as compared with the status at the Baseline visit. The 0-5 rating scale was used: 0: cleared, 1: much improved, 2: minimally improved, 3: unchanged, 4: minimally worse and 5: much worse; where higher score indicates worse condition and lower score indicates clear toenail.
Time Frame: Week 52
Population: ITT analysis set. All participants were available at the time of assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Albaconazole 400 mg (36 Weeks) Oral Weekly | Albaconazole 400 mg (24 Weeks) Oral Weekly | Albaconazole 200 mg (36 Weeks) Oral Weekly | Albaconazole 100 mg (36 Weeks) Oral Weekly | Placebo
Number analyzed (Participants) | 116 | 117 | 117 | 117 | 115
Percentage of participants | 71 [62.4 to 79.0] | 62 [53.6 to 71.2] | 61 [51.8 to 69.5] | 45 [36.3 to 54.3] | 10 [4.2 to 14.9]
Statistical Analysis 1: Comparison: Albaconazole 400 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Albaconazole 400 mg (24 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Albaconazole 200 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Albaconazole 100 mg (36 Weeks) Oral Weekly vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAE) and AEs were collected throughout the study (approximately up to Week 62). SAEs were reported for 62 weeks and non-SAEs reported for treatment period only (36 weeks).
Description: ITT analysis set was used for reporting AE and SAE. The datasets for adverse events could not be located to generate separate non-SAE table.
Arm/Group | Albaconazole 400 mg (36 Weeks) Oral Weekly | Albaconazole 400 mg (24 Weeks) Oral Weekly | Albaconazole 200 mg (36 Weeks) Oral Weekly | Albaconazole 100 mg (36 Weeks) Oral Weekly | Placebo
All-Cause Mortality (participants affected / at risk) | 0/116 | 1/117 | 0/117 | 1/117 | 0/115
Serious Adverse Events (participants affected / at risk) | 4/116 | 7/117 | 3/117 | 6/117 | 2/115
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albaconazole 400 mg (36 Weeks) Oral Weekly (N=116) | Albaconazole 400 mg (24 Weeks) Oral Weekly (N=117) | Albaconazole 200 mg (36 Weeks) Oral Weekly (N=117) | Albaconazole 100 mg (36 Weeks) Oral Weekly (N=117) | Placebo (N=115)
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Peripartum cardiomyopathy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.